CLINICAL TRIAL: NCT02029378
Title: Inhibition of Complement Activation (Eculizumab) in Guillain-Barre Syndrome Study
Acronym: ICA-GBS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GN12NE462
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-09-23 (Estimated); Status verified 2014-09

CONDITIONS: Gullian Barre Syndrome
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eculizumab (Experimental): Eculizumab, 900 mg intravenously once a week
  Interventions: Drug: Eculizumab
- Placebo (Placebo Comparator): Matched placebo, intravenously once a week

INTERVENTIONS:
Drug: Eculizumab
  Arms: Eculizumab

SUMMARY:
Guillian-Barre Syndrome (GBS) is the most frequent cause of acute neuromuscular weakness in the Western World and can occur at any age. GBS is a rpadily progressive 'inflammatory' disorder of the perihperal nerves often leading to sever paresis of the limbs. Most GBS patients also have sensory disturbances (tingling or dull feeling) and pain. Some patients also have double vision or problems with swallowing. GBS mau also involve the respiratory muscles, leading to insufficient ventilation and admission to an intensive care unit. GBS pateints have a vairable prognosis; 20-30% require mechnical ventilation for a period ranging from weeks to months, 20% are unable to walk after 6 months nad 3-5% dies. Progression of weakness in GBS is usually rapid and reaches its peak within 4 weeks in the majority of patients, but many develop their maximum deficit within 2 weeks. Thereafter, the patients have a variable prognosis.

GBS is a treatable disorder. Intravenous immunoglobulin (IVIg) 2g/kg administered in 5 days was shown to be effective when administered within the first two weeks after onset of symptoms, and is considered the treatment of choice by most experts in the field. Although the standard treatment for GBS is a single course of IVIg (2g/kg administered in 5 days), many patients fails to recover abd remain with substantial disability. Patients with GBS and especially those with a poor prognosis potentially may benefit from more powerful abd when possible a more mechanistically rational therapy.

Recent experimental evidence suggests that complement activation palys a crucial role in the development of neuromuscular weakness in GBS making complement inhibitors and regulators attracive therapeutic targets. Our hypothesis is that Eculizumab, with its function as a complement inhibitor, will be very effective in preventing progression of weakness in patients with GBS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years diagnosed with GBS according to NINDS diagnostic criteria
* Onset of weakness due to GBS is less than 2 weeks ago
* Patients who are unable to walk unaided for >10 metres (grade >3 on GBS disability scale)
* Patients who are being considered for or already on IVIg treatment
* First dose of eculizumab must be started within 2 weeks from onset of weakness and any time during the IVIg treatment period
* Signed informed consent

Exclusion Criteria:

* Age <18 years
* Patients who are being considered for, or already on, plasma exchange
* Pregnancy or lactation
* Patients show clear clinical evidence of a polyneuropahty caused by e.g. diabetes mellitus (except mild sensory), alcoholism, severe vitamin deficiency, and porphyria
* Patients received immunosuppressive treatment (e.g. azathioprine, cyclosporine, mycofenolatemofetil, tacrolimus, sirolimus or > 20 mg prednisolone daily) during the last month
* Patients known to have severe concurrent disease, like malignancy, severe cardiovascular disease, AIDS, severe COPD, TB
* Inability to comply with study related procedures or appointments during 6 months
* Any condition that in the opinion of the investigator could increase the patient's risk by participating in the study or confound the outcome of the study
* Related to the administration of eculizumab:

Unresoled Neisseria meningitidisinfection of history of meningococcal infection Unsuitable for antibiotic prophylaxis (e.g due to allergy) Known hypersensitivity to eculizumab, murine proteins or to any of the excipients Known or suspected hereditary complement deficiencies Women of child-bearing potential who are unwilling to use effective contraception during treatment and for 5 months after treatment is completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Determine the incidence of AE/SAEs after treatment with eculizumab and IVIg compared to placebo controls | 6 months
  Primary safety endpoint
Improvement of one or more grade in functional outcome (on the 6 point GBS disability scale) at 4 weeks | 4 weeks
  Primary efficacy endpoint

SECONDARY OUTCOMES:
Ability to walk unaided (GBS disability score 2) at 8 weeks | 8 weeks
Time taken to improve by at least one grade (on the GBS disability scale) | 8 weeks
Time taken to walk independently | 1 year
Difference in GBS disability score at maximum disability completed with 6 months | 6 months
Percentage of patients with a clinically relevant improvement in R-ODS score | 6 months
  An increase from Baseline in R-ODS score by at least 6 points on the centile metric score at 4 weeks and 6 months
Percentage of patients with a clinically relevant improvement in ONLS | 6 months
  Defined as an increase from baseline in ONLS score by at least 1 point at 4 weeks and 6 months
Requirement for ventilatory support (GBS disability score 5) | 4 weeks
Duration of ventilatory support | 8 weeks
Occurrence of relapse | 2 years
Dearth within the first 6 months | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Southern General Hospital, Glasgow, United Kingdom

REFERENCES:
- [Derived] Davidson AI, Halstead SK, Goodfellow JA, Chavada G, Mallik A, Overell J, Lunn MP, McConnachie A, van Doorn P, Willison HJ. Inhibition of complement in Guillain-Barre syndrome: the ICA-GBS study. J Peripher Nerv Syst. 2017 Mar;22(1):4-12. doi: 10.1111/jns.12194. PMID 27801990